CLINICAL TRIAL: NCT01436097
Title: Financial Incentives for Healthy Eating: A Randomized Pilot Study
Brief Title: Randomized Trial of Healthy Eating Interventions
Acronym: WTE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Scott Halpern, Assistant Professor of Medicine (Pulmonary & Critical Care) and Epidemiology Deputy Director, Center for Health Incentives and Behavioral Economics, University of Pennsylvania
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: WTE-814279; RC2AG036592 (NIH)
Record Dates: First submitted 2011-09-14; First posted 2011-09-19 (Estimated); Last update posted 2013-01-15 (Estimated); Status verified 2013-01

CONDITIONS: Nutrition Therapy
Keywords: Healthy Eating; Health Behavior; Incentive; Work-site
MeSH Terms: conditions — Health Behavior

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Usual Care arm (Active Comparator): Participants will have access through the Way to Health portal to web-based educational materials and recipes related to healthy eating. They will be informed they will receive up to $50 in reimbursements for completing the surveys that are part of the Way To Eat program as follows: $20 for completing the intake questionnaire and weigh-in and $30 reimbursements for completing the exit questionnaire and weigh-in.
  Interventions: Behavioral: Usual Care
- Information provision intervention (Experimental): Participants in the Information provision group will receive the same care as those in the Usual Care arm. In addition, the Information provision group participants will receive weekly reminders about the benefits of eating five servings of fruits and vegetables a day and their Way to Health portal will provide graphical depictions of their produce purchase proportions through information from their Price Plus card. This data will be available to them throughout the entire intervention.
  Interventions: Behavioral: Information provision intervention
- Information provision + flat incentive (Experimental): Participants assigned to the Information provision + flat group will earn back 15% of what they spent on groceries for the week if they spend at least 15% of their total grocery budget on fresh produce in addition to receiving the same treatment as the Information provision arm.
  Interventions: Behavioral: information provision + flat incentive
- Information provision + tiered incentive (Experimental): In addition to receiving all features of the Information provision treatment the participants assigned to the Information provision + tiered incentive group would earn back increasing percentages of their grocery spending for meeting increasing targets of produce consumption. In this arm, the more participants spend on produce the more money they can earn back.
  Interventions: Behavioral: Information provision + tiered incentive

INTERVENTIONS:
Behavioral: Information provision intervention — Participant will have access to weekly data showing how much produce they are purchasing. No incentives will be given under this arm. They will also receiving information on weekly purchases, online resources, and weekly reminders on eating healthy.
  Arms: Information provision intervention
Behavioral: information provision + flat incentive — Participants will earn back 15% of what they spent on groceries for the week if they spend at least 15% of their total grocery budget on fresh produce in addition to receiving the same treatment as the IP arm. They will also receiving information on weekly purchases, online resources, and weekly reminders on eating healthy.
  Arms: Information provision + flat incentive
Behavioral: Information provision + tiered incentive — In addition to receiving information on weekly purchases, online resources, and weekly reminders on eating healthy the participants assigned to the IP + tiered incentive group would earn back increasing percentages of their grocery spending for meeting increasing targets of produce consumption.
  Arms: Information provision + tiered incentive
Behavioral: Usual Care — Participants will have access through the Way to Health portal to web-based educational materials and recipes related to healthy eating. They will be informed they will receive up to $50 in reimbursements for completing the surveys that are part of the Way To Eat program as follows: $20 for completing the intake questionnaire and weigh-in and $30 reimbursements for completing the exit questionnaire and weigh-in.
  Arms: Usual Care arm

SUMMARY:
Interventions to increase the consumption of fruits and vegetables to date have shown promise, but many have limited public health impact due to the lack of scalability of their designs. The investigators propose to examine the effectiveness and feasibility of an intervention for promoting increased consumption of fruits and vegetables by incentivizing their purchase. Collaborating with UpLift Solutions, the investigators will enroll shoppers in this Randomized Clinical Trial using the research infrastructure called the Way to Health platform. (called the Way to Health platform, and approved as a Prime protocol by the IRB as reference # 811860).

Hypothesis: providing patients with financial incentives can promote healthier behaviors (e.g.: eating healthier).

DETAILED DESCRIPTION:
This is a pilot study under the IRB-approved umbrella protocol number 811698 named Penn-CMU Roybal Center on Behavioral Economics and Health. Interventions to increase the consumption of fruits and vegetables to date have shown promise, but many have limited public health impact due to the lack of scalability of their designs. Many interventions only provided information on what constitutes healthier eating or provided discounts on specific products.Other interventions were limited in generalizability due to utilization of very specific eating establishments or vending machines.By contrast, the investigators propose to examine the effectiveness and feasibility of an intervention for promoting increased consumption of fruits and vegetables by incentivizing their purchase where the overwhelming majority of food is sold: grocery stores. Collaborating with Brown's Super Stores and UpLift Solutions leadership, the investigators will enroll shoppers in this Randomized Clinical Trial using our the web-based research infrastructure called the Way to Health platform.

The primary aim of this project is to generate preliminary evidence of the efficacy of two financial incentive structures in promoting the allocation of a greater percentage of ones grocery budget to the purchase of fresh fruits and vegetables (hereafter, produce). Secondary aims are to evaluate these interventions effects on (1) self-reported consumption of produce, and (2) weight. Salutary goals of this pilot study are to document feasibility of using Price Plus cards for incentive studies, and to expand the functionality of the Way Health platform.

ELIGIBILITY:
Inclusion Criteria:

* Current Parkside Brown's Super Stores shoppers who use a Price Plus Card
* Have regular internet access
* Spend at least $30 per household member per week on groceries
* Spend 10% or less of their grocery budget on produce
* 18 years of age or older
* weekly grocery shoppers

Exclusion Criteria:

* Plan to move in the next 4 months
* Plan to stop shopping at Brown's Super Stores in the next 4 months
* Plan to stop using their Price Plus card in the next 4 months
* Receive any assistance like SNAP or WIC

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2011-10; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Changes from baseline in proportion of fruit and vegetable purchases | weekly for 3 months
  Changes from baseline in proportion of grocery money that is spent on fruits and vegetables each week for 12 weeks across each intervention group. Fruits and vegetables, or produce, will be defined by the food product itself, not its location in the store. Produce in this study will include frozen and canned fruits and vegetables as well as fresh fruits and vegetables.

SECONDARY OUTCOMES:
Changes from baseline in self-reported consumption of fruits and vegetables | weekly for 3 months
  Changes from baseline in self-reported consumption of fruits and vegetables each week for 12 weeks across each intervention.
Changes in body weight from baseline to end of treatment (12 weeks after intervention start) | Baseline and an average of 12-14 weeks after intervention start
  Changes in body weight from baseline to end of treatment (12 weeks after intervention start; pre- and post- intervention).

CONTACTS AND LOCATIONS:
Overall Officials: Scott D Halpern, MD, Ph.D., Principal Investigator — University of Pennsylvania; Kathryn A Saulsgiver, MS, PhD, Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Background] Appel LJ, Moore TJ, Obarzanek E, Vollmer WM, Svetkey LP, Sacks FM, Bray GA, Vogt TM, Cutler JA, Windhauser MM, Lin PH, Karanja N. A clinical trial of the effects of dietary patterns on blood pressure. DASH Collaborative Research Group. N Engl J Med. 1997 Apr 17;336(16):1117-24. doi: 10.1056/NEJM199704173361601. PMID 9099655
- [Background] Lin, B. Diet Quality Usually Varies by Income Status. Washington, DC: U.S. Department of Agriculture, Economic Research Service. Amber Wave, 3(5), 2005.
- [Background] Morland K, Wing S, Diez Roux A, Poole C. Neighborhood characteristics associated with the location of food stores and food service places. Am J Prev Med. 2002 Jan;22(1):23-9. doi: 10.1016/s0749-3797(01)00403-2. PMID 11777675
- [Background] Blisard, N & Stewart, H. Food Spending in American Households, 2003-04. Economic Information Bulletin 59033, United States Department of Agriculture, Economic Research Service 2007.
- [Result] Blair SN, Jacobs DR Jr, Powell KE. Relationships between exercise or physical activity and other health behaviors. Public Health Rep. 1985 Mar-Apr;100(2):172-80. PMID 3920715
- [Result] Coulson NS, Eiser C, Eiser JR. Diet, smoking and exercise: interrelationships between adolescent health behaviours. Child Care Health Dev. 1997 May;23(3):207-16. doi: 10.1111/j.1365-2214.1997.tb00964.x. PMID 9158910
- [Result] Basiotis, PP, Carlson, A, Gerrior, SA, Juan, WY, & Lino, M. Nutrition Insight 28: Report Card on the Quality of Americans' Diets. Family Economics and Nutrition Review 16(2): 66-68, 2004.
- [Result] Garasky, S, Morton, LW, & Greder, K. The Food Environment and Food Insecurity: Perceptions of Rural, Suburban, and Urban Food Pantry Clients in Iowa. Family Economics and Nutrition Review 16(2): 41-48, 2004.
- [Result] Seymour JD, Yaroch AL, Serdula M, Blanck HM, Khan LK. Impact of nutrition environmental interventions on point-of-purchase behavior in adults: a review. Prev Med. 2004 Sep;39 Suppl 2:S108-36. doi: 10.1016/j.ypmed.2004.04.002. PMID 15313080
- [Result] Kristal AR, Goldenhar L, Muldoon J, Morton RF. Evaluation of a supermarket intervention to increase consumption of fruits and vegetables. Am J Health Promot. 1997 Jul-Aug;11(6):422-5. doi: 10.4278/0890-1171-11.6.422. PMID 10168262
- [Result] French SA, Wechsler H. School-based research and initiatives: fruit and vegetable environment, policy, and pricing workshop. Prev Med. 2004 Sep;39 Suppl 2:S101-7. doi: 10.1016/j.ypmed.2003.10.007. PMID 15313079
- [Result] Glanz K, Hoelscher D. Increasing fruit and vegetable intake by changing environments, policy and pricing: restaurant-based research, strategies, and recommendations. Prev Med. 2004 Sep;39 Suppl 2:S88-93. doi: 10.1016/j.ypmed.2004.03.002. PMID 15313077
- [Result] French SA, Jeffery RW, Story M, Breitlow KK, Baxter JS, Hannan P, Snyder MP. Pricing and promotion effects on low-fat vending snack purchases: the CHIPS Study. Am J Public Health. 2001 Jan;91(1):112-7. doi: 10.2105/ajph.91.1.112. PMID 11189801
- [Result] Basiotis, PP, Carlson, A, Gerrior, SA, Juan, WY, & Lino, M. The Healthy Eating Index: 1999-2000. U.S. Department of Agriculture, Center for Nutrition Policy and Promotion. CNPP-12, 2002
- [Result] Lin, BH, Yen, ST, Dong, D, & Smallwood, DM. Economic incentives for dietary improvement among food stamp recipients. Contemporary Economic Policy 28 (4): 524-536, 2010
- [Result] He FJ, Nowson CA, Lucas M, MacGregor GA. Increased consumption of fruit and vegetables is related to a reduced risk of coronary heart disease: meta-analysis of cohort studies. J Hum Hypertens. 2007 Sep;21(9):717-28. doi: 10.1038/sj.jhh.1002212. Epub 2007 Apr 19. PMID 17443205
- [Result] Mann J, Aune D. Can specific fruits and vegetables prevent diabetes? BMJ. 2010 Aug 18;341:c4395. doi: 10.1136/bmj.c4395. No abstract available. PMID 20724401
- [Result] Brown L, Rimm EB, Seddon JM, Giovannucci EL, Chasan-Taber L, Spiegelman D, Willett WC, Hankinson SE. A prospective study of carotenoid intake and risk of cataract extraction in US men. Am J Clin Nutr. 1999 Oct;70(4):517-24. doi: 10.1093/ajcn/70.4.517. PMID 10500021
- [Result] Christen WG, Liu S, Schaumberg DA, Buring JE. Fruit and vegetable intake and the risk of cataract in women. Am J Clin Nutr. 2005 Jun;81(6):1417-22. doi: 10.1093/ajcn/81.6.1417. PMID 15941896
- [Result] Drewnowski A. The cost of US foods as related to their nutritive value. Am J Clin Nutr. 2010 Nov;92(5):1181-8. doi: 10.3945/ajcn.2010.29300. Epub 2010 Aug 18. PMID 20720258
- [Result] Halpern SD, Karlawish JH, Casarett D, Berlin JA, Asch DA. Empirical assessment of whether moderate payments are undue or unjust inducements for participation in clinical trials. Arch Intern Med. 2004 Apr 12;164(7):801-3. doi: 10.1001/archinte.164.7.801. PMID 15078651
- [Result] Halpern SD, Raz A, Kohn R, Rey M, Asch DA, Reese P. Regulated payments for living kidney donation: an empirical assessment of the ethical concerns. Ann Intern Med. 2010 Mar 16;152(6):358-65. doi: 10.7326/0003-4819-152-6-201003160-00005. PMID 20231566